CLINICAL TRIAL: NCT02053883
Title: A Phase II/III, Double-Blind, Randomized, Placebo-Controlled, Multicenter Study to Assess the Efficacy and Safety of Cethrin in Subjects With Acute Cervical Spinal Cord Injury
Brief Title: Cethrin in Acute Cervical Spinal Cord Injury
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Compound recently partnered with another company for continued development.
Sponsor: BioAxone BioSciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BA-210-201
Record Dates: First submitted 2014-01-31; First posted 2014-02-04 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Spinal Cord Injury
Keywords: SCI; spinal cord injury; biologic drug; rho; paralysis; paraplegia; tetraplegia; quadriplegia; trauma; central nervous system; fibrin sealant; neurosurgery; cervical; regeneration; neurotrauma
MeSH Terms: conditions — Spinal Cord Injuries; Night Blindness, Congenital Stationary, Autosomal Dominant 1; Paralysis; Paraplegia; Quadriplegia; Wounds and Injuries | interventions — exoenzyme C3, Clostridium botulinum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Placebo (Placebo Comparator): Fibrin sealant only.
  Interventions: Drug: Placebo
- Cethrin (BA-210) - Low Dose (Experimental): Low dose of Cethrin in a fibrin sealant.
  Interventions: Drug: Cethrin (BA-210)
- Cethrin (BA-210) - High Dose (Experimental): High dose of Cethrin in a fibrin sealant.
  Interventions: Drug: Cethrin (BA-210)

INTERVENTIONS:
Drug: Cethrin (BA-210) — High or low doses of Cethrin administered extradurally in a fibrin sealant during spinal decompression/stabilization surgery.
  Arms: Cethrin (BA-210) - High Dose; Cethrin (BA-210) - Low Dose
Drug: Placebo — Fibrin sealant alone administered extradurally during spinal decompression/stabilization surgery.
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled Phase IIb/III study designed to evaluate the efficacy and safety of Cethrin as a treatment for acute cervical spinal cord injury. During the trial, high and low doses of Cethrin will be compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, ages 18-62, inclusive
* Acute cervical spinal cord injury at a neurological level of C4-C6
* AIS Grade A or B
* Scheduled to undergo decompression/stabilization surgery within five days of injury
* Written or verbal consent from patient or legally authorized representative that patient is able and willing to comply with the study protocol, including follow-up visits

Exclusion Criteria:

* Participation in any other clinical trial for acute SCI, including previous Cethrin trial
* Inability to receive study medication within five days of injury
* Acute SCI from gunshot or penetrating/stab wound; peripheral nerve injury; brachial plexus injury; complete spinal cord transection; or multifocal SCI
* Significant hemorrhage on MRI/CT scan
* Females who are breastfeeding or have a positive serum pregnancy test
* Body mass index (BMI) of ≥ 35 kg/m2 at screening
* History of an adverse reaction to a fibrin sealant or its human or bovine components
* Use of intravenous heparin in previous 48 hours, aspirin-containing products in previous 24 hours, thrombolytics in previous 12 hours
* Hemophilia or other bleeding abnormality (platelet level lower than 100 X 109/L, activated partial thromboplastin time or international normalized ratio higher than the upper limit of normal, or baseline hematocrit lower than 0.25)
* Unconsciousness or other impairment that precludes reliable ASIA examination
* Known immunodeficiency, including human immunodeficiency virus, or use of immunosuppressive or cancer chemotherapeutic drugs
* Clinically significant pre-existing neurological, cardiac, respiratory, hepatic, or renal disease

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
American Spinal Injury Association (ASIA) Upper Extremity Motor Score Recovery | Baseline to 6 Months

SECONDARY OUTCOMES:
ASIA Total Motor Score Recovery | Baseline to 6 Months
ASIA Impairment Scale (AIS) Grade Recovery | Baseline to 6 Months
Motor Neurological Level Recovery | Baseline to 6 Months
ASIA Sensory Score Recovery | Baseline to 6 Months
Spinal Cord Independence Measure (SCIM) III (Total Score, Self-Care Subscore) | 6 Months
Graded Redefined Assessment of Strength, Sensibility and Prehension (GRASSP) | 6 Months
Incidence of Adverse Events | 0-6 Months